CLINICAL TRIAL: NCT05756634
Title: Health and Wellness After Preterm Birth: Randomized Controlled Trial of Enhanced Support After Preterm Birth
Brief Title: Health and Wellness After Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-019198; K23HD102560 (NIH)
Record Dates: First submitted 2023-02-20; First posted 2023-03-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Preterm Birth; Health Care Utilization; Tobacco Use; Contraceptive Usage; Depression; Weight, Birth
Keywords: Preconception Care; Interconception care; Postpartum care; Preventive health care; Care coordination; Motivational Interviewing
MeSH Terms: conditions — Premature Birth; Patient Acceptance of Health Care; Tobacco Use; Contraception Behavior; Depression; Birth Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCAPB (intervention) (Experimental): Intervention participants will receive an intervention focused on health care navigation and motivational enhancement.
  Interventions: Behavioral: Care Coordination after Preterm Birth (CCAPB)
- Usual Care (Placebo Comparator): Usual care participants will not receive the intervention.
  Interventions: Behavioral: Care Coordination after Preterm Birth (CCAPB)

INTERVENTIONS:
Behavioral: Care Coordination after Preterm Birth (CCAPB) — For participants randomized to CCAPB, the care coordinator will follow a manualized intervention to support care planning, health care access, and wellbeing. Contact with participants will be initiated as soon as possible after enrollment, and will continue until six months after enrollment.

SUMMARY:
This study continues an adaptation of the behavioral intervention Care Coordination After Preterm Birth (CCAPB). This is a pragmatic pilot randomized controlled feasibility trial of CCAPB with baseline and post-intervention assessments.

DETAILED DESCRIPTION:
Interventionists will be trained in care coordination strategies and Motivational Interviewing (MI) techniques. Following training, investigators will enroll eligible women from a postpartum unit at a single hospital, or within 4 weeks of birth.The primary outcome of this study is acceptability and feasibility of the intervention and study procedures as measured by the Acceptability of Intervention Measure, participant completion of study data collection, and interventionist completion of planned intervention modules.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 14 - 45
* History of preterm birth (< 34 weeks gestational age or 34 - 36 weeks with identifiable risk factors for recurrent preterm birth which may including: low preventive care utilization, tobacco use, obesity, depression or anxiety, history of unmet contraceptive needs, chronic or pregnancy-associated hypertension or diabetes. )
* Intention to seek pediatric care at one of two pediatric primary care sites
* Medicaid insurance

Exclusion Criteria:

* History of sterilization procedure.
* Plan to move away from the area or transfer pediatric primary care within six months of enrollment.
* Limited English proficiency.
* History of organ failure or malignancies.

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of the CCAPB intervention | up to 6 months
  Investigators will use the Acceptability of Intervention Measure (modified) with a threshold of > 3 indicating acceptability.

SECONDARY OUTCOMES:
Patient reported stress. | up to 6 months
  Stress will be measured by the validated Perceived Stress Scale (PSS).The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful.Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Sleep-related impairment | up to 6 months
  Sleep-related impairment will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment - Short Form 8a.
  The Sleep-Related Impairment instrument is a self-reported tool used to document perceived overall sleep-related impairment (or sleep-wake function) over the past seven days. The PROMIS method of scoring uses responses to each item for each participant. For most PROMIS instruments, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population.
Depression symptoms | up to 6 months
  Depression symptoms will be measured by the Edinburgh Postnatal Depression Scale (EPDS). The 10-question Edinburgh Postnatal Depression Scale (EPDS) is used to identify patients at risk for perinatal depression. Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity.
Autonomous motivation | up to 6 months
  Autonomous motivation will be measured using the Autonomous Motivation and External Regulation scales of the Treatment Self-Regulation Questionnaire (10 items, range 7 - 70, Cronbach alpha 0.90). This is a self administered questionnaire with a higher score indicating higher emotion regulation strategy.
Completion of recommended postpartum care | up to 6 months
  Completion of recommended postpartum care will be assessed by patient health record review.
Contraceptive Use | up to 6 months
  Contraceptive Use will be measured using an item from the self administered PRAMS questionnaire.
  Are you or your husband or partner doing anything now to keep from getting pregnant? No / Yes (if Yes proceed to next)
  What kind of birth control are you or your husband using now to keep from getting pregnant?
  PRAMS is an ongoing, site-specific, population-based surveillance system designed to identify groups of women and infants at high risk for health problems, to monitor changes in health status, and to measure progress towards goals in improving the health of mothers and infants.
Tobacco use | up to 1 month
  Tobacco use will be assessed by asking participants "Have you smoked any cigarettes in the past 30 days?"
Multivitamin use | up to 6 months
  Multivitamin use will be assessed by asking participants "Are you currently taking a multivitamin?"
Autonomy Support | up to 6 months
  Autonomy support will be measured with the self regulated short form of the Health Care Climate Questionnaire (6 items, range 6 - 42, Cronbach alpha 0.82). Scores on the short form 6-item version are calculated by averaging the individual item scores. Higher average scores represent a higher level of perceived autonomy support.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Gregory, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will be used to refine the protocol for further testing. There are no plans to share individual participant data.